CLINICAL TRIAL: NCT02137447
Title: A Prospective Observational Study of the Use of Negative Pressure Wound in High Risk Surgical Closed Incisions.
Brief Title: Use of Negative Pressure Wound Therapy in High Risk Surgical Closed Incisions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel Dante Yeh, Trauma and Critical Care Attending Surgeon, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P002484
Record Dates: First submitted 2014-05-08; First posted 2014-05-13 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: High Risk Abdominal Wounds
Keywords: Prevena; faster healing time; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Negative Pressure Wound Therapy (Experimental): After the completion of the operation, incisional skin closure was performed using sutures or staples and the wound was then covered with the Negative Pressure Wound therapy Prevena Incision Management System (Kinetic Concepts Inc) as per the manufacturer's instructions of use. Continuous negative pressure was applied at 125 mm Hg.
  For inpatients, wounds were assessed every 48 hours by inspection and palpation. The dressing was not routinely removed, but the surrounding skin was assessed for cellulitis. The NPWT dressing was removed between post-operative day 5 and 7
  Interventions: Device: Negative Pressure treatment

INTERVENTIONS:
Device: Negative Pressure treatment

SUMMARY:
The purpose of this study is to investigate the use of Negative Pressure Wound Therapy in high risk surgical wounds to evaluate the rate of surgical site infections (SSIs).

Hypothesis:

Historically, the average rates of infective complications in surgical wounds types are 7.7% in clean wounds, 15% for contaminated and 35-40% for dirty wounds. The application of Prevena ™ Incision Management System (Kinetic Concepts Inc, San Antonio, TX) is expected to reduce these rates by 50%.

DETAILED DESCRIPTION:
Wound infections continue to be a common and costly problem after surgery. Surgical site infections (SSIs) are the second most common type of health care - associated infections (HAI), occurring in 2% to 5% of patients undergoing surgery in the United States. This percentage corresponds to approximately 300,000 to 500,000 surgical site infections (SSIs) estimated to occur each year.

Most SSIs that do not involve implants are diagnosed within 3 weeks post--operatively . SSIs lead to increased hospital stay, cost, and risk of death. The cost attributable to SSI range from $3,000 to $29,000 per SSI per patient depending on the type of operation; thus, the total annual cost approximately reaches the $10 billions. On other analyses documented nearly 1 million additional inpatient-days and $1.6 billion in excess costs , as well as up to twice the costs of a patient without SSI. Moreover, SSIs increase mortality risk by 2 to 11 fold 11, while the 77% of deaths in patients with SSI are attributed directly to the SSIs. Several organizations have put forth guidelines for definition and recommendations to decrease their incidence. Attempts have been made to stratify patients into various categories on the basis of the type of surgical procedure and risk factors the patients have, including diabetes, malnutrition, and hypoxemia. These systems have been used to develop criteria for the prevention of wound infection.

Appropriate timing and dosing of antibiotics, type of skin preparation, temperature of the patient in the operating room, blood oxygen level of the patient during surgery, and management of blood glucose levels all have been standardized in an attempt to decrease wound infection rates . In addition, debridement of all tissue that may contribute to wound infection, particularly ischemic skin and subcutaneous tissue, is standard surgical procedure. Standardization has led to a small decrease in incidence but has not led to a significant reduction in the overall rate. One reason for this is the multifactorial nature of SSI development. Factors regarding patients and pre-operative status, operative procedures and intra-operative events, as well as postoperative course, all need to be addressed, and there is not a complete understanding of their range and impact. What is known is that at the time of wound closure, one needs a minimal number of bacteria in the wound, and the wound itself must be reasonably well perfused and oxygenated. After surgery, wound perfusion and oxygenation are evaluated by clinical appearance. If the wound does not appear ischemic, it is assumed that perfusion and oxygenation are adequate. Unfortunately, this has never been quantified. Negative-pressure wound therapy (NPWT) has been used to speed the healing of open wounds.

How this occurs is not completely understood, but increased generation of granulation tissue at the margins of the open wound implies increased generation of blood vessels and substances needed to promote wound healing.

The theory of negative pressure is the stimulation of wound healing on the basis of improved perfusion to the wound. This has been seen in open wounds and has recently been applied to closed surgical wounds thought to be at high risk for infection. Negative-pressure wound therapy was also applied to closed wounds in an attempt to improve wound perfusion and oxygenation, which in theory would eliminate these two variables from the wound infection equation.

Techniques - Procedures Complete closure of the abdominal wall and skin follows the completion of the index surgical procedure. Closed suction drains may be used at the time of skin closure in any patient who requires skin flap elevation to attain skin closure. Skin closure will be accomplished with dermal sutures and / or staples. Wound coverage will be done with the NPWT Prevena ™ Incision Management System (Kinetic Concepts Inc, San Antonio, TX). The application of the NPWT will be done as per manufacturer's instructions of use. The application of continuous negative pressure will be applied at 125 mm Hg.Antibiotics will be given to all patients. The post-operative use of antibiotics in the clear contaminated and contaminated cases will be 24-hour of prophylactic administration. The post-operative use of antibiotics for the dirty (infected) cases will be of therapeutic administration, as clinically indicated. In infected patients, cultures will be taken at the time of the index procedure, and the antibiotic treatment will be targeted to the culture results. Wounds will be assessed every 48 hours by dressing changes, and also at the time of final dressing removal and at 2 and 4 weeks after surgery. The dressing removal will take place at discharge OR at 5 - 7 post-operative days OR if clinically indicated, whichever comes first. Post-discharge follow-up The patients will be followed-up per routine at the surgical clinic. At 2 and 4 weeks after the date of the operation a formal evaluation will take place. Both evaluations must be in person at the surgical clinic.

ELIGIBILITY:
Inclusion Criteria:

* All five of the following criteria must be present for enrollment into the study:

  1. Signed written informed consent must be provided by the patient or by patient's legally acceptable representative, if patient unable to consent.
  2. Age > 18 years
  3. Abdominal operation entering the peritoneal cavity under general anesthesia for colostomy or ileostomy reversal or enterocutaneous fistula excision
  4. Clean - contaminated OR contaminated OR dirty wound (as defined by Wound Infection Surveillance) OR use of skin flaps for skin closure.
  5. Complete closure of the surgical wound including the skin.

Exclusion Criteria:

* 1) Known allergic reaction at the wound dressing parts of the Prevena ™ Incision Management System.

(Included but not limited to: sensitivity to silver, allergic or hypersensitivity reaction to acrylic adhesives).

2) Inability to close the abdominal wall at the index procedure. 3) Inability to close the skin at the index procedure. 4) Patients under 18 years old. 5) Pregnant women test

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Negative Pressure treatment
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infections Within 1 Month (4 Weeks ) From Index Operation
Description: Incidence of SSIs within 1 month (4 weeks) from the index operation. SSI is defined by the Centers for Disease Control and Prevention's National Healthcare Surveillance Network
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group: Negative Pressure Wound Therapy (NPWT) to closed surgical incision
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Participants | 1

2. Secondary Outcome: Composite Secondary Outcomes of Non-infectious Abdominal Wound Complications, Damage to the Skin Caused by the Dressing, Need to End the Treatment Prior to Discharge or Prior to 5-7 Post-operative Days, and Need for Reapplication of the System.
Description: Secondary (composite) outcomes:
  1. other non infectious abdominal wound complications,
  2. damage to the skin caused by the dressing
  3. need to end the treatment prior the discharge OR prior to 5 -7 post- operative days.
  4. need for re-application of the system for any reason
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10)
death (General disorders) | 1 (1) — death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10)
urinary tract infection (Renal and urinary disorders) | 1 (1)
intra-abdominal abscess requiring percutaneous drainage (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No